CLINICAL TRIAL: NCT02691416
Title: Role of Propofol Postconditioning on Oxidative Stress and Cognitive Function in Patients Undergoing Intracranial Aneurysm Surgery.
Brief Title: Role of Propofol Postconditioning on Oxidative Stress and Cognitive Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Third Central Clinical College of Tianjin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ThirdCCCTianjin
Record Dates: First submitted 2016-02-03; First posted 2016-02-25 (Estimated); Results first posted 2016-09-02 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2016-02

CONDITIONS: Cerebral Arterial Aneurysm
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol postconditioning (Experimental): 1.2mg/L propofol
  Interventions: Drug: propofol postconditioning; Drug: sevoflurane
- sevoflurane (Experimental): 0.5%-2% sevoflurane
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: propofol postconditioning — administrated Target Controlled Infusion(TCI) of propofol (Cp 1.2ug/ml) and decreased sevoflurane with a Bispectral index (BIS) value of 40-60 to maintain anesthesia after clamp removal
  Arms: propofol postconditioning
Drug: sevoflurane — 0.5%-2% sevoflurane with BIS 40-60

SUMMARY:
The purpose of this study was to evaluate differences between propofol postconditioning and sevoflurane anesthesia in the intracranial aneurysm surgery about antioxidant effect.

DETAILED DESCRIPTION:
intracranial aneurysm surgery may lead to regional ischemic reperfusion injury. Propofol, as an antioxidative phenol, has been demonstrated that mitigate the brain I/R in rats.

As for sevoflurane, some investigation indicated that sevoflurane is able to reduce oxidative stress in cell(except neuronal cell lines ) and rodent models, but the antioxidant effect did not found in human minor incision surgeries, furthermore, oxidative stress was raised in the major surgeries including orthopedic surgeries, hysterectomy, cholecystectomy, and thoracotomy

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis intracranial aneurysm surgery ,
* American Society of Anesthesiologists (ASA)Ⅰ-Ⅱ.

Exclusion Criteria:

* severe hepatic and renal dysfunction
* coagulation disorder
* taking antioxidant perioperative period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haiyun Wang, Study Director — The Third Central Clinical College of Tianjin Medical University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2014 to January 2016, patients who were undergoing intracranial aneurysm surgery at hospital and consistent with the criterion of American Society of Anesthesiologists (ASA)Ⅰ-Ⅱ,but without severe hepatic and renal dysfunction, coagulation disorder were recruited.
Groups:
- Propofol Postconditioning: Group propofol postconditioning was administrated TCI of propofol (Cp 1.2ug/ml) and decreased sevoflurane concentration with a BIS value of 40-60 to maintain anesthesia after clamp removal immediately.
Period: Overall Study
Arm/Group | Propofol Postconditioning | Sevoflurane
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propofol Postconditioning: 1.2ug/ml propofol Group propofol postconditioning was administrated TCI of propofol (Cp 1.2ug/ml) and decreased sevoflurane concentration with a BIS value of 40-60 to maintain anesthesia after clamp removal immediately.
- Total: Total of all reporting groups
Arm/Group | Propofol Postconditioning | Sevoflurane | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Evidences of Clinically Definite Oxidative Stress Confirmed by ELISA Kit
Description: Evidences of clinically definite oxidative stress :Superoxide dismutase activity, Hydroxyl radical
Time Frame: before induction,after clamping removal ,operation ending ,1,3,7days post surgery
Measure: Mean (Standard Deviation); unit: U/ml
Groups:
- Propofol Postconditioning: 1.2ug/ml propofol
  propofol: Group propofol postconditioning was administrated TCI of propofol (Cp 1.2ug/ml) and decreased sevoflurane concentration with a BIS value of 40-60 to maintain anesthesia after clamp removal immediately.
Arm/Group | Propofol Postconditioning | Sevoflurane
Number analyzed (Participants) | 30 | 30
U/ml
  Superoxide dismutase activity of before induction | 72.87 (23.15) | 74.02 (21.27)
  Superoxide dismutase activity of clamping removal | 67.10 (16.52) | 65.91 (16.07)
  Superoxide dismutase activity of operation ending | 66.74 (16.50) | 51.58 (14.92)
  Superoxide dismutase activity of 1days postsurgery | 66.80 (16.56) | 52.82 (14.93)
  Superoxide dismutase activity of 3days postsurgery | 69.27 (16.66) | 57.35 (17.36)
  Superoxide dismutase activity of 7days postsurgery | 69.02 (16.95) | 59.33 (17.30)
  Hydroxyl radical of before induction | 5.30 (6.46) | 6.60 (6.49)
  Hydroxyl radical of clamping removal | 15.80 (4.42) | 16.22 (5.23)
  Hydroxyl radical of operation ending | 12.54 (4.32) | 15.29 (5.30)
  Hydroxyl radical of 1days post surgery | 10.32 (4.61) | 13.65 (5.37)
  Hydroxyl radical of 3days post surgery | 8.05 (4.80) | 12.46 (5.33)
  Hydroxyl radical of 7days post surgery | 6.33 (5.57) | 10.32 (5.16)

2. Primary Outcome: Evidences of Clinically Definite Oxidative Stress Confirmed by ELISA
Description: Evidences of clinically definite oxidative stress:8-isoprostane,as a reliable biomarkers of lipid peroxidation
Time Frame: before induction, after clamping removal,operation ending,1,3,7days post surgery
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Propofol Postconditioning | Sevoflurane
Number analyzed (Participants) | 30 | 30
pg/ml
  8-isoprostane of before induction | 1.15 (0.14) | 1.18 (0.14)
  8-isoprostane of clamping removal | 1.19 (0.15) | 1.22 (0.14)
  8-isoprostane of operation ending | 1.54 (0.16) | 1.70 (0.18)
  8-isoprostane of 1days post surgery | 1.51 (0.16) | 1.64 (0.21)
  8-isoprostane of 3days post surgery | 1.48 (0.17) | 1.60 (0.18)
  8-isoprostane of 7days post surgery | 1.38 (0.18) | 1.49 (0.19)

3. Primary Outcome: Evidences of Clinically Definite Oxidative Stress:Micronuclei
Description: Evidences of clinically definite oxidative stress:micronuclei confirmed by Cytokinesis-block Micronucleus Test
Time Frame: before induction,clamping removal ,operation ending,1,3,7days post surgery
Measure: Mean (Standard Deviation); unit: number of micronuclei/1000 BN cells
Arm/Group | Propofol Postconditioning | Sevoflurane
Number analyzed (Participants) | 30 | 30
number of micronuclei/1000 BN cells
  micronuclei of before induction | 185.83 (21.69) | 186.40 (19.87)
  micronuclei of clamping removal | 194.57 (25.27) | 195.73 (24.21)
  micronuclei of operation ending | 230.77 (25.00) | 375.87 (30.90)
  micronuclei of 1days post surgery | 278.73 (30.86) | 402.27 (27.60)
  micronuclei of 3days post surgery | 248.43 (30.88) | 338.00 (30.85)
  micronuclei of 7days post surgery | 201.33 (28.98) | 243.63 (29.59)

4. Primary Outcome: Evidences of Clinically Definite Oxidative Stress Confirmed by High Performance Liquid Chromatography
Description: Evidences of clinically definite oxidative stress :α- tocopherol,γ- tocopherol which was used to assess the antioxidant defense.
Time Frame: before induction,after clamping removal ,operation ending ,1,3,7days post surgery
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Propofol Postconditioning | Sevoflurane
Number analyzed (Participants) | 30 | 30
ug/ml
  α- tocopherol of before induction | 12.67 (1.96) | 12.22 (1.83)
  α- tocopherol of clamping removal | 6.13 (1.81) | 6.12 (1.68)
  α- tocopherol of opertaion ending | 6.71 (1.79) | 5.91 (1.68)
  α- tocopherol of 1days post surgery | 8.97 (1.87) | 8.23 (1.51)
  α- tocopherol of 3days post surgery | 10.02 (2.06) | 9.31 (1.56)
  α- tocopherol of 7days post surgery | 11.54 (1.84) | 10.98 (1.80)
  γ- tocopherol of before induction | 0.52 (0.08) | 0.53 (0.08)
  γ- tocopherol of clamping removal | 0.59 (0.09) | 0.57 (0.09)
  γ- tocopherol of opertaion ending | 0.84 (0.10) | 0.75 (0.10)
  γ- tocopherol of 1days post surgery | 0.76 (0.11) | 0.69 (0.10)
  γ- tocopherol of 3days post surgery | 0.70 (0.13) | 0.62 (0.09)
  γ- tocopherol of 7days post surgery | 0.68 (0.13) | 0.60 (0.11)

5. Primary Outcome: Evidences of Clinically Definite Oxidative Stress: Nuclear Buds
Description: Evidences of clinically definite oxidative stress:nuclear buds Confirmed by Cytokinesis-block Micronucleus Test
Time Frame: before induction,clamping removal ,operation ending,1,3,7days post surgery
Measure: Mean (Standard Deviation); unit: number of nuclear buds/1000 BN cells
Arm/Group | Propofol Postconditioning | Sevoflurane
Number analyzed (Participants) | 30 | 30
number of nuclear buds/1000 BN cells
  nuclear buds of before induction | 50.40 (8.84) | 53.93 (9.11)
  nuclear buds of clamp ing removal | 54.33 (8.56) | 57.43 (8.44)
  nuclear buds of operation ending | 61.10 (9.16) | 62.87 (10.47)
  nuclear buds of 1days post surgery | 62.73 (10.38) | 65.07 (11.27)
  nuclear buds of 3days post surgery | 58.00 (8.31) | 61.70 (10.03)
  nuclear buds of 7days post surgery | 54.87 (9.56) | 55.67 (11.49)

6. Primary Outcome: Evidences of Clinically Definite Oxidative Stress: Nucleoplasmic Bridges
Description: Evidences of clinically definite oxidative stress: nucleoplasmic bridges confirmed by Cytokinesis-block Micronucleus Test
Time Frame: before induction,clamping removal ,operation ending,1,3,7days post surgery
Measure: Mean (Standard Deviation); unit: number of nucleoplasmic bridges/1000 BN
Groups:
- Propofol Postconditioning: 1.2ug/mL propofol
  propofol:Group propofol postconditioning was administrated TCI of propofol (Cp 1.2ug/ml) and decreased sevoflurane concentration with a BIS value of 40-60 to maintain anesthesia after clamp removal immediately
Arm/Group | Propofol Postconditioning | Sevoflurane
Number analyzed (Participants) | 30 | 30
number of nucleoplasmic bridges/1000 BN
  nucleoplasmic bridges of before induction | 66.50 (9.92) | 68.73 (8.22)
  nucleoplasmic bridges of clamp ing removal | 78.77 (13.66) | 80.80 (12.34)
  nucleoplasmic bridges of operation ending | 88.40 (14.08) | 96.23 (12.70)
  nucleoplasmic bridges of 1days post surgery | 96.83 (14.74) | 111.93 (11.77)
  nucleoplasmic bridges of 3days post surgery | 86.87 (11.29) | 96.37 (12.70)
  nucleoplasmic bridges of 7days post surgery | 79.20 (11.17) | 87.83 (12.85)

7. Secondary Outcome: Mini Mental State Examination (MMSE)
Description: A questionnaires is used to assess the cognitive function of patients in clinical,the total range was 0-30,and 27-30 were considered as normal value,<27 were considered as recognitive dysfunction.
Time Frame: before induction,1,3,7days post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Propofol Postconditioning: 1.2ug/mL propofol
  propofol: Group propofol postconditioning was administrated TCI of propofol (Cp 1.2ug/ml) and decreased sevoflurane concentration with a BIS value of 40-60 to maintain anesthesia after clamp removal
Arm/Group | Propofol Postconditioning | Sevoflurane
Number analyzed (Participants) | 30 | 30
units on a scale
  before induction of MMSE | 27.63 (1.43) | 27.23 (1.63)
  1days post surgery of MMSE | 23.40 (1.87) | 17.73 (2.02)
  3 days post surgery of MMSE | 24.43 (2.18) | 20.33 (1.94)
  7 days post surgery of MMSE | 27.00 (2.00) | 24.30 (1.97)

8. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: as for outcome 7
Time Frame: before induction,1,3,7days post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propofol Postconditioning | Sevoflurane
Number analyzed (Participants) | 30 | 30
units on a scale
  before induction of MoCA | 20.43 (2.39) | 19.87 (2.60)
  1days post surgery | 21.53 (2.58) | 19.20 (2.31)
  3days post surgery | 22.53 (2.68) | 20.80 (2.73)
  7days post surgery | 26.20 (2.27) | 23.10 (2.73)

ADVERSE EVENTS:
Time Frame: 7days
Arm/Group | Propofol Postconditioning | Sevoflurane
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No